CLINICAL TRIAL: NCT00895531
Title: Comparison of Peripheral Nerve Blocks vs. Combination of Peripheral Nerve Block and DepoDur in Total Knee Joint Replacement: A Prospective, Randomized Study
Brief Title: Combination of Peripheral Nerve Block and DepoDur in Total Knee Joint Replacement
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: University of Louisville (Other)
Collaborators: EKR Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.0255
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Knee Replacement, Total; Morphine
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peripheral Nerve group (Active Comparator): Group will receive sciatic catheter placed before or after surgery by subgluteal approach with the use of ultrasound. The ischial tuberosity will be identified with the ultrasound probe and its midpoint marked. A catheter will be inserted and placed perineurally. If placed preoperatively, the catheter will be flushed with normal saline or 5% dextrose and will not be dosed until after surgery. After the patient is in the PACU and the surgeons have verified the sciatic nerve function, the sciatic catheter will be dosed with 35 mL 0.25% ropivacaine.
  Interventions: Procedure: sciatic nerve block
- Depodur Group (Experimental): patients will have an L2-L3 epidural placed while they are in the sitting position before or after femoral catheter placement. They will receive 7.5 mg Depodur via the epidural catheter. All of these patients will receive Singular 10 mg and Claritin 10 mg before the epidural Depodur is placed, as per our protocol of patients receiving EREM.
  Interventions: Drug: Depodur

INTERVENTIONS:
Drug: Depodur — 7.5 mg Depodur via the epidural catheter
  Other Names: morphine sulfate extended-release liposome injection
  Arms: Depodur Group
Procedure: sciatic nerve block — The sciatic nerve will be identified at the subgluteal level with ultrasound. A point 3 cm lateral and 4 cm caudad will be marked. Patients will be placed in the lateral position. A 18 G Tuohy needle will be inserted at a 45° angle until a peroneal or tibial twitch is obtained at 1.5 mA. Once the current can be reduced to obtain a twitch less than 0.5 mA, a catheter will be inserted and placed perineurally. If placed preoperatively, the catheter will be flushed with normal saline or 5% dextrose and will not be dosed until after surgery. After the patient is in the PACU and the surgeons have verified the sciatic nerve function, the sciatic catheter will be dosed with 35 mL 0.25% ropivacaine.
  Other Names: Nerve block, sciatic
  Arms: Peripheral Nerve group

SUMMARY:
The investigators hypothesize that patients who receive a femoral catheter with low dose epidural Depodur will experience comparable or superior pain relief than those who receive both femoral and sciatic catheters. In addition, the investigators hypothesize that the one catheter will be less time consuming to place and facilitate early ambulation of the patient.

DETAILED DESCRIPTION:
After obtaining written informed consent, all patients will be sedated with 1-5 mg midazolam and up to 100 mcg fentanyl before any procedure is performed. They will be attached to standard ASA monitors and their vital signs recorded before sedation and every 5 minutes throughout the procedure. They will receive supplemental oxygen 2-4 LPM with a nasal canula. They will be given 1 g acetaminophen orally with a sip of water before sedation.

The randomization envelope will be opened and the patient will be randomized to one of the two groups.

All patients will receive a femoral nerve block after identification of the landmarks or with ultrasound guidance and a femoral catheter will be inserted perineurally. The patients will be placed supine position for the procedure. The femoral artery will be identified either by ultrasound or a hand held Doppler. A point 1 cm lateral to the femoral artery and 1 cm below the inguinal crease is marked. A 5 cm Tuohy needle (Pajunk Medical) will be inserted at a 45° angle at 1.5 mA and 1 Hz. Once a brisk quadriceps twitch is identified, the needle will be positioned accurately so as to establish quadriceps stimulation at ≤ 0.5 mA.

The peripheral nerve catheter will be inserted through the needle. Once the catheter is positioned satisfactorily in the perineural area, it will be tunneled subcutaneously and a sterile dressing will be applied to cover the catheter completely. Ropivacaine (30 mL of 0.5%) will be injected through the catheter after frequent aspirations. The block will be assessed by sensory and motor assessments at 5, 10, 15, and 30 minutes. Sensory testing will be performed on the anterior aspect of the knee (femoral nerve), medial aspect of the knee (obturator nerve) and the lateral aspect of the thigh (lateral femoral cutaneous nerve). The block will be considered complete when no cold discrimination was observed (Score 2), partial when cold discrimination was decreased (score 1), and absent when normal cold discrimination was observed (Score 0). Femoral motor block will also be assessed during the same period by testing knee extension, and will be considered complete when no extension is observed, partial when quadriceps motor force is decreased and absent when normal quadriceps function is observed. Patients with complete sensory block of the femoral and obturator nerves after 15 minutes will be included in the study.

Group I: Peripheral Nerve group: This group will have a sciatic catheter placed either before or after surgery. They will receive a sciatic catheter by subgluteal approach with the use of ultrasound. The ischial tuberosity will be identified with the ultrasound probe and its midpoint marked. A point 3 cm lateral and 4 cm caudad will be marked. Patients will be placed in the lateral position. A 18 G Tuohy needle will be inserted at a 45° angle until a peroneal or tibial twitch is obtained at 1.5 mA. Once the current can be reduced to obtain a twitch less than 0.5 mA, a catheter will be inserted and placed perineurally. If placed preoperatively, the catheter will be flushed with normal saline or 5% dextrose and will not be dosed until after surgery. After the patient is in the PACU and the surgeons have verified the sciatic nerve function, the sciatic catheter will be dosed with 35 mL 0.25% ropivacaine.

Group II: Depodur Group: Preoperatively this group of patients will have an L2-L3 epidural placed while they are in the sitting position before or after femoral catheter placement. They will receive 7.5 mg Depodur via the epidural catheter. All of these patients will receive Singular 10 mg and Claritin 10 mg before the epidural Depodur is placed, as per our protocol of patients receiving EREM.

All patients will receive general anesthesia with fentanyl 2 mcg/kg, ketamine 0.2 mg/kg, and propofol, as needed, for induction of anesthesia. The patients will be paralyzed with succinylcholine, rocuronium, or any other non-depolarizing muscle relaxant of choice of anesthesiologist. Analgesia will be maintained at the discretion of the anesthesiologist overseeing the case. Anesthesia will be maintained with a volatile anesthetic and oxygen or TIVA to maintain BIS between 40 and 50. Vital signs will be recorded every 15 minutes. They will also receive dexamethasone 4 mg, metoclopramide 20 mg IV at induction and ondansetron 4 mg after induction, if they have more than 40% risk of PONV as per their Apfel score.

Patients will be extubated at the end of the case and transferred to PACU. If patients complain of pain, they will receive fentanyl 25-50-mcg increments as per the discretion of PACU nurse to achieve a VRS < 4. Patients may be prescribed a morphine PCA (1 mg morphine with a 6-minute lockout) for postoperative pain relief in the PACU once their pain is stable at VRS<4.

All patients will be prescribed acetaminophen 1000 mg every 6 hours for 3 days after surgery. They will be prescribed metoclopramide 20 mg IV PRN every 6 hours as rescue medication for nausea and/or vomiting for 2 days postoperatively. Patients still nauseous will get Promethazine (Phenergan) 6.25-12.5 mg as second line rescue.

Once the patients are transported to the floor, they will be monitored with continuous pulse-oximetry for the first 48 hours. Other vital signs (Pulse, NIBP and Respiratory Rate) will be monitored every hour for the first 12 hours, every 2 hrs from 12-24 hours, and every 4 hours from 24 to 48 hours (ASA 2009 Guidelines for neuraxial opioids).

Postoperative knee joint rehabilitation will involve continuous passive motion (CPM) of the knee joint twice a day. The physical therapist will be asked to record the VRS on movement and the range of motion after placement of the CPM machine.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for total knee replacement or revision of total knee replacement
* Agree to have a regional technique including neuraxial analgesia for post-operative analgesia
* Be 18 to 70 years old
* Classified as ASA score I-III

Exclusion Criteria:

* Allergic to morphine
* Allergic to local anesthetics
* Been on opioids for more than 4 weeks
* Not willing to be randomized
* On anticoagulation medications that prevent placement of epidural
* Sensitive to effects of neuraxial opioids
* BMI>35
* Severe COPD
* Obstructive sleep apnea (OSA, see below). Each patient will be asked the questions below to determine their risk for OSA (STOP questionnaire). Patients who answer yes to 3 or more of the major criteria of the STOP questionnaire and have one of the minor criteria will be excluded from the study

STOP Questionnaire for OSA

Major Criteria:

S- Do you snore loudly (louder than talking or loud enough to be heard through closed doors)?

T-"Do you often feel tired, fatigued, or sleepy during daytime?

O-"Has anyone observed you stop breathing during your sleep?

P-"Do you have or are you being treated for high blood pressure?

Minor Criteria:

* BMI>35
* Age>50 yrs
* Neck Circumference>40 cm
* Male gender

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anupama Wadhwa, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peripheral Nerve Group | Depodur Group
Started | 38 | 37
Completed | 38 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peripheral Nerve Group | Depodur Group | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 37 | 75
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 32 | 28 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain
Description: Pain as reported on a verbal rating scale ( VRS) (0-10, 0 = no pain, 10 = worse pain imaginable).
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peripheral Nerve Group | Depodur Group
Number analyzed (Participants) | 38 | 37
units on a scale | 5 (3) | 6 (2)
Statistical Analysis 1: Comparison: Peripheral Nerve Group vs Depodur Group; Test type: Superiority; p = 0.95, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Peripheral Nerve Group | Depodur Group
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/37
Other Adverse Events (participants affected / at risk) | 0/38 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peripheral Nerve Group (N=38) | Depodur Group (N=37)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes